CLINICAL TRIAL: NCT01313767
Title: A Randomized, Double Blind, Multi-center, Active Drug Controlled Clinical Trial to Compare the Efficacy and Safety of MEDITOXIN® Versus BOTOX® in Treatment of Post Stroke Upper Limb Spasticity
Brief Title: MEDITOXIN® Versus BOTOX® in the Treatment of Post-stroke Spasticity of the Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-PRT-ST01
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Spasticity
Keywords: spasticity; upperlimb; Botulinum toxin
MeSH Terms: conditions — Muscle Spasticity | interventions — Botulinum Toxins, Type A; 3-deoxyglycero-galacto-nonulosonic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meditoxin® (Experimental): Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A
- Botox® (Active Comparator): Botulinum Toxin type A
  Interventions: Drug: Botulinum Toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A
  Other Names: Neuronox®, Siax®
  Arms: Meditoxin®
Drug: Botulinum Toxin type A — Botulinum Toxin type A
  Other Names: Botox®
  Arms: Botox®

SUMMARY:
This study is a randomized, double blind, multi-center, active drug controlled, phase III clinical trial to compare the efficacy and safety of MEDITOXIN® versus BOTOX® in treatment of post stroke upper limb(wrist, finger, thumb) spasticity

Approximately 196 subjects(1:1 group ratio)will be enrolled. Subjects will receive a single treatment of intramuscular Investigational product up to 360U. The subjects will be observed every 4 weeks until 12 weeks post injection. Outcome measures include Modified Ashworth Scale (MAS), Disability Assessment Scale (DAS), Global Assessment Scale(patient or caregiver/investigator) and Carer burden scale. The primary efficacy endpoint is the change from baseline at week 4 for wrist flexor muscle tone as measured on the Modified Ashworth Scale. Safety parameters will also be measured including adverse events, vital signs and clinical laboratory tests (haematology, serum chemistry and urinanalysis).

DETAILED DESCRIPTION:
Each completed subject will attend 4~5 clinic visits. The maximum study duration is 15 weeks. Only one upper limb (eligible inclusion/exclusion criteria) will be injected and evaluated in the study. Maximun injection dose is 360U.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 20 years
2. ≥ 6 weeks since the last stroke
3. ≥ 2 points in the focal spasticity of wrist flexor and ≥ 1 points at least one of elbow flexor and finger flexor as measured on MAS(0 to 4)
4. Targeted one functional disability item (i.e., hygiene, dressing, pain, or cosmesis) with a rating of 2 or greater on DAS (0 to 3)
5. Informed consent has been obtained.

Exclusion Criteria:

1. Neuromuscular disorders such as Lambert-Eaton syndrome, myasthenia gravis, or amyotrophic lateral sclerosis
2. History(within 6 months of screening visit) or planned(during study period) treatment with phenol or alcohol injection or surgery in the target limb
3. History(within 6 months of screening visit) or planned(during study period) treatment with tendon lengthening in the target limb
4. Fixed joint/muscle contracture
5. Severe atrophy
6. Concurrent treatment with an intrathecal baclofen
7. History(within 3 months of screening visit) Planned(during study period) treatment with Botulinum Toxin
8. Known allergy or sensitivity to study medication or its components
9. Concurrent or planed Muscle relaxants and/or benzodiazepine medication

   * If patient has taken these medication stable from one month before screening and no treatment changes are not planned during the study, participation is allowed.
10. Current Physical, occupational, Splinting therapy

    * If these therapy regimens will be permitted if they has been stable in the one month before screening;no treatment and no changes are planned during the study.
11. Patient who are participating in other clinical trials at the screening
12. Females who are pregnant, breatfeeding,or planning a pregnancy during the study period, or female of childbearing potential, not using a reliable means of centraception.
13. Patients who are not eligible for this study at the discretion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moon Suk Bang, Ph.D, Principal Investigator — Seoul National Universtiy Hospital, 101 Daehak-ro Jong-gu, Seoul 110-744, Korea; Min Ho Chun, Ph.D, Principal Investigator — Asan Medical Center, 388-1 Pungnap-2 dong, Songpa-Gu, Seoul, 138-736, Korea; Nam Jong Baik, Ph. D, Principal Investigator — University Bundang Hospital, Seoul National Univ. Bundang Hospital, Gumi-dong, Bundang-gu, Seongnam-si, Gyeonggi-do, Korea; Si Uk Lee, Ph.D, Principal Investigator — SMG-SNU Boramae Medical Center, 41, Borame-Gill, Dong Gjak-Gu, Seoul, 156-707, Seoul, Korea; Beom Seon Gwon, Ph.D, Principal Investigator — Dongguk University International Hospital, Siksa-dong, Ilsandong-gu, Goyang-si, Gyeonggi-do, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo HG, Paik NJ, Lee SU, Oh BM, Chun MH, Kwon BS, Bang MS. Neuronox versus BOTOX in the Treatment of Post-Stroke Upper Limb Spasticity: A Multicenter Randomized Controlled Trial. PLoS One. 2015 Jun 1;10(6):e0128633. doi: 10.1371/journal.pone.0128633. eCollection 2015. PMID 26030192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, total 208 patients were screened and total 196 subjects (98 subjects per group) were randomized, except 12 screening-failures, at 5 study sites.
Pre-assignment Details: Total 9 subjects were prematurely discontinued from the study due to unmet inclusion/exclusion criteria found after randomization, AEs/SAEs, consent withdrawal and follow-up lost: 7 subjects in study group (7.14%) and 2 subjects in control group (2.04%). Thus total 187 subjects (91 in study group; 96 in control group) completed the study.
Groups:
- Meditoxin®; Botox®: Clostridium Botulinum toxin type A, up to total 360U injected into selected sites, Intra-muscle
Period: Overall Study
Arm/Group | Meditoxin® | Botox®
Started | 98 | 98
Completed | 91 | 96
Not Completed | 7 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | Meditoxin® | Botox® | Total
Number analyzed (Participants) | 94 | 98 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 69 | 136
  >=65 years | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.54 (11.03) | 56.99 (13.01) | 57.26 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 65 | 67 | 132
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 94 | 98 | 192
Weight [Mean (Standard Deviation); unit: kg] | 65.51 (10.27) | 62.94 (9.67) | 64.18 (10.02)

OUTCOME MEASURES:

1. Primary Outcome: MAS(Modified Ashworth Scale) of Wrist Flexor
Description: Change from baseline at week 4 for wrist flexor muscle tone as measured on the MAS(Modified Ashworth Scale). The Modified Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Baseline and 4 weeks
Population: The analysis was performed on the Full Analysis Set population which consisted of 94 subjects receiving Meditoxin and 98 subjects for Botox.
Measure: Mean (Standard Deviation); unit: Scores on a MAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 94 | 98
Scores on a MAS Scale
  Baseline | 2.41 (0.61) | 2.52 (0.66)
  Week 4 | 1.02 (0.81) | 0.96 (0.64)
  Change(Week4-Baseline) | -1.39 (0.79) | -1.56 (0.81)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; The difference between the two groups was provided with 95% CI. If the upper limit of CI is no greater than 0.45 (non-inferiority margin), the study group was determined not inferior to the control group. Additionally, difference between groups in change from baseline to week 4 in wrist flexor MAS score was compared using two sample t-test; Test type: Non-Inferiority or Equivalence — 90% of the power, 0.45 of non-inferiority margin; p = 0.1347, t-test, 2 sided; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.05 to 0.40]

2. Secondary Outcome: MAS(Modified Ashworth Scale) of Wrist Flexor
Description: Change from baseline at week 8 and 12 for wrist flexor muscle tone as measured on the MAS(Modified Ashworth Scale).
  The Modified Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Baseline, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 94 subjects receiving Meditoxin and 98 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a MAS scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 94 | 98
Scores on a MAS scale
  Baseline | 2.41 (0.61) | 2.52 (0.66)
  Week 8 | 1.07 (0.78) | 1.04 (1.16)
  Week 12 | 1.16 (0.86) | 1.16 (0.66)
  Change(Week 8 - Baseline) | -1.35 (0.77) | -1.48 (0.87)
  Change(Week12 - Baseline) | -1.25 (0.78) | -1.36 (0.84)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in wrist flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.2591, t-test, 2 sided; Mean Difference (Final Values) = 0.07
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in wrist flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.3395, t-test, 2 sided; Mean Difference (Final Values) = 0.09

3. Secondary Outcome: MAS(Modified Ashworth Score) of Elbow Flexor
Description: Change from baseline at week 4, week 8 and 12 for elbow flexor muscle tone as measured on the MAS(Modified Ashworth Scale).
  The Modified Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 87 subjects receiving Meditoxin and 94 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a MAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 87 | 94
Scores on a MAS Scale
  Baseline | 2.33 (0.75) | 2.18 (0.65)
  Week 4 | 1.26 (0.73) | 1.30 (0.58)
  Week 8 | 1.36 (0.54) | 1.41 (0.58)
  Week 12 | 1.45 (0.68) | 1.52 (0.60)
  Change(Week 4 - Baseline) | -1.07 (0.73) | -0.87 (0.71)
  Change(Week 8 - Baseline) | -0.97 (0.74) | -0.77 (0.72)
  Change(Week 12 - Baseline) | -0.88 (0.75) | -0.65 (0.74)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in elbow flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.0675, t-test, 2 sided; Mean Difference (Final Values) = -0.2
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in elbow flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.0605, t-test, 2 sided; Mean Difference (Final Values) = -0.2
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in elbow flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.0429, t-test, 2 sided; Mean Difference (Final Values) = -0.23

4. Secondary Outcome: MAS(Modified Ashworth Score) of Finger Flexor
Description: Change from baseline at week 4, week 8 and 12 for finger flexor muscle tone as measured on the MAS(Modified Ashworth Scale).
  The Modified Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 82 subjects receiving Meditoxin and 83 Botox.
Measure: Mean (Standard Deviation); unit: Score on a MAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 82 | 83
Score on a MAS Scale
  Baseline | 2.37 (0.80) | 2.48 (0.75)
  Week 4 | 1.01 (0.67) | 1.05 (0.66)
  Week 8 | 1.15 (0.62) | 1.17 (0.66)
  Week 12 | 1.20 (0.68) | 1.30 (0.66)
  Change(Week 4 - Baseline) | -1.36 (0.90) | -1.42 (0.94)
  Change(Week 8 - Baseline) | -1.23 (0.89) | -1.30 (0.91)
  Change(Week 12 - Baseline) | -1.18 (0.90) | -1.16 (0.91)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in finger flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.6954, t-test, 2 sided; Mean Difference (Final Values) = 0.06
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in finger flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.6024, t-test, 2 sided; Mean Difference (Final Values) = 0.07
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in finger flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.9316, t-test, 2 sided; Mean Difference (Final Values) = -0.02

5. Secondary Outcome: MAS(Modified Ashworth Score) of Thumb Flexor
Description: Change from baseline at week 4, 8, 12 for thumb flexor muscle tone as measured on MAS.
  The Modified Ashworth Scale is a well known and commonly used scale in clinical trials with spasticity. It was considered to be the best clinical tool for measuring resistance to movement. It was used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 54 subjects receiving Meditoxin and 58 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a MAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 54 | 58
Scores on a MAS Scale
  Baseline | 1.94 (0.73) | 1.94 (0.74)
  Week 4 | 0.89 (0.71) | 0.69 (0.66)
  Week 8 | 1.01 (0.67) | 0.84 (0.77)
  Week 12 | 1.06 (0.84) | 0.96 (0.69)
  Change(Week 4 - Baseline) | -1.06 (0.85) | -1.25 (0.83)
  Change(Week 8 - Baseline) | -0.94 (0.85) | -1.09 (0.85)
  Change(Week 12 - Baseline) | -0.89 (0.99) | -0.98 (0.86)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in thumb flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.2284, t-test, 2 sided; Mean Difference (Final Values) = 0.19
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in thumb flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.3221, t-test, 2 sided; Mean Difference (Final Values) = 0.15
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in thumb flexor MAS score was compared using two sample t-test; Test type: Superiority or Other; p = 0.5930, t-test, 2 sided; Mean Difference (Final Values) = 0.09

6. Secondary Outcome: Improvement Rate on the MAS(Modified Ashworth Score) of Wrist Flexor
Description: Improvement in the injected site muscle tone at week 4, 8 and 12 as measured by MAS(Modified Ashworth Score) of wrist flexor.
  * A treatment response is defined as 1-point improvement on the MAS(Modified Ashworth Score) of injection site.
Time Frame: week 4, week 8, week 12
Population: as for outcome 2
Measure: Number; unit: Subjects who improved 1-point on MAS
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 94 | 98
Subjects who improved 1-point on MAS
  Week 4 | 77 | 88
  Week 8 | 77 | 80
  Week 12 | 71 | 77
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 4 from baseline in wrist flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.1585, Chi-squared; Risk Difference (RD) = -0.07
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 8 from baseline in wrist flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.9596, Chi-squared; Risk Difference (RD) = 0.0028
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 12 from baseline in wrist flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.6164, Chi-squared; Risk Difference (RD) = -0.0304

7. Secondary Outcome: Improvement Rate on the MAS(Modified Ashworth Score) of Elbow Flexor
Description: Improvement in the injected site muscle tone at week 4, 8 and 12 as measured by MAS(Modified Ashworth Score) of elbow flexor.
  * A treatment response is defined as 1-point improvement on the MAS(Modified Ashworth Score) of injection site
Time Frame: week 4, week 8, week 12
Population: as for outcome 3
Measure: Number; unit: Subjects who improved 1-point on MAS
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 87 | 94
Subjects who improved 1-point on MAS
  Week 4 | 56 | 52
  Week 8 | 49 | 42
  Week 12 | 46 | 39
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 4 from baseline in elbow flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.1802, Chi-squared; Risk Difference (RD) = 0.0980
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 8 from baseline in elbow flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.1176, Chi-squared; Risk Difference (RD) = 0.1164
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 12 from baseline in elbow flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.1252, Chi-squared; Risk Difference (RD) = 0.1138

8. Secondary Outcome: Improvement Rate on the MAS(Modified Ashworth Score) of Finger Flexor
Description: Improvement in the injected site muscle tone at week 4, 8 and 12 as measured by MAS(Modified Ashworth Score) of finger flexor.
  * A treatment response is defined as 1-point improvement on the MAS(Modified Ashworth Score) of injection site.
Time Frame: week 4, week 8, week 12
Population: as for outcome 4
Measure: Number; unit: Subjects who improved 1-point on MAS
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 82 | 83
Subjects who improved 1-point on MAS
  Week 4 | 58 | 64
  Week 8 | 51 | 60
  Week 12 | 47 | 54
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 4 from baseline in finger flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.3431, Chi-squared; Risk Difference (RD) = 0.0980
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 8 from baseline in finger flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.1329, Chi-squared; Risk Difference (RD) = -0.1097
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 12 from baseline in finger flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.2611, Chi-squared; Risk Difference (RD) = 0.0853

9. Secondary Outcome: Improvement Rate on the MAS(Modified Ashworth Score) of Thumb Flexor
Description: Improvement in the injected site muscle tone at week 4, 8 and 12 as measured by MAS(Modified Ashworth Score) of thumb flexor.
  * A treatment response is defined as 1-point improvement on the MAS(Modified Ashworth Score) of injection site.
Time Frame: week 4, week 8, week 12
Population: as for outcome 5
Measure: Number; unit: Subjects who improved 1-point on MAS
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 54 | 58
Subjects who improved 1-point on MAS
  Week 4 | 34 | 41
  Week 8 | 28 | 37
  Week 12 | 27 | 30
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 4 from baseline in thumb flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.4623, Chi-squared; Risk Difference (RD) = -0.0654
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 8 from baseline in thumb flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.2007, Chi-squared; Risk Difference (RD) = -0.1194
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency of responders who have improved at least 1-point on the MAS at week 12 from baseline in thumb flexor was compared using Pearson's chi-square test; Test type: Superiority or Other; p = 0.8553, Chi-squared; Risk Difference (RD) = 0.0172

10. Secondary Outcome: DAS(Disability Assessment Scale) of Hygiene
Description: Change From Baseline to week 4, 8, 12 in the DAS(Disability Assessment Scale) for the Principal Therapeutic Target as Hygiene.
  The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 39 subjects receiving Meditoxin and 34 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a DAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 39 | 34
Scores on a DAS Scale
  Baseline | 2.62 (0.49) | 2.74 (0.45)
  Week 4 | 1.90 (1.02) | 2.09 (0.87)
  Week 8 | 1.85 (0.99) | 2.12 (0.88)
  Week 12 | 1.87 (0.98) | 2.12 (0.84)
  Change(Week 4 - Baseline) | -0.72 (0.79) | -0.65 (0.65)
  Change(Week 8 - Baseline) | -0.77 (0.67) | -0.62 (0.65)
  Change(Week 12 - Baseline) | -0.74 (0.75) | -0.62 (0.60)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in DAS score of hygiene was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.6040, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.07
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in DAS score of hygiene was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.3233, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.15
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in DAS score of hygiene was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.4469, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.12

11. Secondary Outcome: DAS(Disability Assessment Scale) of Dressing
Description: Change From Baseline to week 4, 8, 12 in the DAS(Disability Assessment Scale) for the Principal Therapeutic Target as Dressing. The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 11 subjects receiving Meditoxin and 15 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a DAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 11 | 15
Scores on a DAS Scale
  Baseline | 2.09 (0.30) | 2.13 (0.35)
  Week 4 | 1.30 (0.67) | 1.07 (0.47)
  Week 8 | 1.36 (0.50) | 1.00 (0.55)
  Week 12 | 1.27 (0.65) | 1.00 (0.55)
  Change(Week 4 - Baseline) | -0.70 (0.67) | -1.07 (0.47)
  Change(Week 8 - Baseline) | -0.73 (0.47) | -1.14 (0.66)
  Change(Week 12 - Baseline) | -0.82 (0.60) | -1.14 (0.66)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in DAS score of dressing was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.1220, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.37
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in DAS score of dressing was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.1016, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.41
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in DAS score of dressing was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.2235, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.32

12. Secondary Outcome: DAS(Disability Assessment Scale) of Limb Position
Description: Change From Baseline to week 4, 8, 12 in the DAS(Disability Assessment Scale) for the Principal Therapeutic Target as Limb Position.
  The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 40 subjects receiving Meditoxin and 47 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a DAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 40 | 47
Scores on a DAS Scale
  Baseline | 2.50 (0.51) | 2.45 (0.50)
  Week 4 | 1.28 (0.55) | 1.29 (0.54)
  Week 8 | 1.27 (0.55) | 1.25 (0.53)
  Week 12 | 1.29 (0.56) | 1.23 (0.47)
  Change(Week 4 - Baseline) | -1.23 (0.62) | -1.15 (0.55)
  Change(Week 8 - Baseline) | -1.23 (0.66) | -1.19 (0.54)
  Change(Week 12 - Baseline) | -1.20 (0.69) | -1.21 (0.55)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in DAS score of limb position was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.5030, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.08
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in DAS score of limb position was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.6934, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.04
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in DAS score of limb position was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.9574, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.01

13. Secondary Outcome: DAS(Disability Assessment Scale) of Pain
Description: Change From Baseline to week 4, 8, 12 in the DAS(Disability Assessment Scale) for the Principal Therapeutic Target as Pain.
  The Disability Assessment Scale consists of the four domains hygiene, dressing, limb position, and pain which were assessed on a 4-point scale with the values 0 (=no disability), 1 (=mild disability), 2 (=moderate disability), and 3 (=severe disability).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 4 subjects receiving Meditoxin and 2 Botox.
Measure: Mean (Standard Deviation); unit: Scores on a DAS Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 4 | 2
Scores on a DAS Scale
  Baseline | 2.00 (0.00) | 2.00 (0.00)
  Week 4 | 1.25 (0.50) | 1.00 (0.00)
  Week 8 | 0.75 (0.50) | 1.00 (0.00)
  Week 12 | 0.50 (0.58) | 0.00 (0.00)
  Change(Week 4 - Baseline) | -0.75 (0.50) | -1.00 (0.00)
  Change(Week 8 - Baseline) | -1.25 (0.50) | -1.00 (0.00)
  Change(Week 12 - Baseline) | -1.50 (0.58) | -2.00 (0.00)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in DAS score of pain was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.7237, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.25
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in DAS score of pain was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.7237, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.25
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in DAS score of pain was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.4017, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.50

14. Secondary Outcome: Global Assessment by Investigator
Description: Global assessment evaluated by investigator at week 12 after injection
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 94 | 98
participants
  Very good | 19 | 19
  Good | 63 | 56
  Moderate | 10 | 18
  Insufficient | 1 | 4
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in frequency distribution of responders on the Global Assessment at week 12 was compared using Fisher's exact test; Test type: Superiority or Other; p = 0.2346, Fisher Exact

15. Secondary Outcome: Global Assessment by Patient or Caregiver
Description: Global assessment evaluated by patient or caregiver at week 12 after injection
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 94 | 98
participants
  Very good | 11 | 10
  Good | 39 | 44
  Moderate | 36 | 35
  Insufficient | 7 | 8
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.9513, Fisher Exact

16. Secondary Outcome: Carer Burden Scale of Cleaning the Palm
Description: The Carer Burden Scale evaluates the impact of antispastic medication on the physical burden of the carer. It was assessed on a 5-point Likert scale which values ranges from 0 (=no difficulty) to 4 (=cannot do the task).
Time Frame: Baseline, week 4, week 8 and week 12
Population: The analysis was performed on the Full Analysis Set population which consisted of 92 subjects receiving Meditoxin and 98 Botox.
Measure: Mean (Standard Deviation); unit: Score on a Carer Burden Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 92 | 98
Score on a Carer Burden Scale
  Baseline | 1.70 (1.16) | 1.67 (1.17)
  Week 4 | 1.26 (1.02) | 1.34 (1.00)
  Week 8 | 1.24 (0.96) | 1.40 (1.09)
  Week 12 | 1.18 (1.05) | 1.44 (1.09)
  Change(Week 4 - Baseline) | -0.40 (1.29) | -0.34 (1.10)
  Change(Week 8 - Baseline) | -0.46 (1.24) | -0.28 (1.09)
  Change(Week 12 - Baseline) | -0.51 (1.34) | -0.23 (1.17)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in carer burden scale of cleaning the palm was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.8088, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.06
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in carer burden scale of cleaning the palm was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.3702, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.18
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in carer burden scale of cleaning the palm was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.1497, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.28

17. Secondary Outcome: Carer Burden Scale of Cutting the Finger-nails
Description: as for outcome 16
Time Frame: Baseline, week 4, week 8 and week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a Carer Burden Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 92 | 98
Scores on a Carer Burden Scale
  Baseline | 2.08 (1.34) | 2.22 (1.27)
  Week 4 | 1.58 (1.30) | 1.89 (1.32)
  Week 8 | 1.57 (1.25) | 1.84 (1.37)
  Week 12 | 1.59 (1.32) | 1.81 (1.35)
  Change(Week 4 - Baseline) | -0.47 (1.26) | -0.34 (1.17)
  Change(Week 8 - Baseline) | -0.51 (1.29) | -0.39 (1.25)
  Change(Week 12 - Baseline) | -0.49 (1.35) | -0.42 (1.19)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in carer burden scale of cutting the finger-nails was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.9634, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.13
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in carer burden scale of cutting the finger-nails was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.7302, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.12
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in carer burden scale of cutting the finger-nails was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.7715, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.07

18. Secondary Outcome: Carer Burden Scale of Putting Shirts on
Description: as for outcome 16
Time Frame: Baseline, week 4, week 8 and week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a Carer Burden Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 92 | 98
Scores on a Carer Burden Scale
  Baseline | 1.79 (1.00) | 1.64 (1.11)
  Week 4 | 1.46 (0.97) | 1.42 (1.10)
  Week 8 | 1.34 (0.96) | 1.28 (0.97)
  Week 12 | 1.32 (1.05) | 1.30 (1.07)
  Change(Week 4 - Baseline) | -0.32 (1.12) | -0.22 (0.98)
  Change(Week 8 - Baseline) | -0.46 (1.11) | -0.37 (1.17)
  Change(Week 12 - Baseline) | -0.48 (1.13) | -0.35 (1.15)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in carer burden scale of putting shirts on was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.9362, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.10
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in carer burden scale of putting shirts on was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.7998, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.09
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in carer burden scale of putting shirts on was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.5436, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.13

19. Secondary Outcome: Carer Burden Scale of Cleaning the Armpit
Description: as for outcome 16
Time Frame: Baseline, week 4, week 8 and week 12
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a Carer Burden Scale
Arm/Group | Meditoxin® | Botox®
Number analyzed (Participants) | 92 | 98
Scores on a Carer Burden Scale
  Baseline | 1.98 (1.21) | 1.97 (1.27)
  Week 4 | 1.56 (1.15) | 1.71 (1.26)
  Week 8 | 1.50 (1.16) | 1.59 (1.29)
  Week 12 | 1.42 (1.15) | 1.69 (1.33)
  Change(Week 4 - Baseline) | -0.39 (1.12) | -0.26 (1.20)
  Change(Week 8 - Baseline) | -0.48 (1.12) | -0.38 (1.26)
  Change(Week 12 - Baseline) | -0.55 (1.19) | -0.28 (1.43)
Statistical Analysis 1: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 4 in carer burden scale of cleaning the armpit was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.7014, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.13
Statistical Analysis 2: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 8 in carer burden scale of cleaning the armpit was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.8884, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.10
Statistical Analysis 3: Comparison: Meditoxin® vs Botox®; Difference between groups in change from baseline to week 12 in carer burden scale of cleaning the armpit was compared using wilcoxon rank sum test; Test type: Superiority or Other; p = 0.2840, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.27

ADVERSE EVENTS:
Time Frame: The subjects were observed every visit after signing an Informed consent form (visit 1) until 12 weeks post injection
Description: All AEs reported during the study period were tabulated and AE incidence was determined.
Arm/Group | Meditoxin® | Botox®
Serious Adverse Events (participants affected / at risk) | 5/98 | 8/98
Other Adverse Events (participants affected / at risk) | 35/98 | 35/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meditoxin® (N=98) | Botox® (N=98)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Behcet's syndrome (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meditoxin® (N=98) | Botox® (N=98)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Consitipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Injection site haematoma (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1) | 3 (5)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Partial seizures (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the results which arise directly or indirectly from the clinical trial in any form shall be the exclusive property of the sponsor.

PIs and the sponsor will discuss, prior to public release of the results, any draft publication or communication made by the investigator. PIs shall not mention any information for a patent or for any intellectual property rights. The sponsor may use or explit all the results at its own discretion, without any limitation to its property right.